CLINICAL TRIAL: NCT01434745
Title: Smith-Lemli Opitz Syndrome: A Clinical Investigation of the Effect of Simvastatin in Patients Receiving Cholesterol Supplementation
Brief Title: SLOS: The Effect of Simvastatin in Patients Receiving Cholesterol Supplementation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment (only one subject enrolled)
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jean-Baptiste Roullet, Clinical Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL073980 (NIH); R01HL073980 (NIH)
Record Dates: First submitted 2011-09-07; First posted 2011-09-15 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: SLOS; Cholesterol Supplementation; Simvastatin
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome | interventions — Simvastatin; Lactose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Lactose
- Simvastatin (Experimental): 0.5 mg/kg body weight/day
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin will be administered as a powder mixed with lactose at the dose of 0.5 mg/kg/day
  Other Names: Zocor, Flolipid
  Arms: Simvastatin
Dietary Supplement: Lactose — Lactose will be administered in a capsule formula.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if simvastatin improves development and behavior in patients with Smith Lemli-Opitz syndrome (SLOS) receiving dietary cholesterol supplementation.

DETAILED DESCRIPTION:
Patients with SLOS receiving dietary cholesterol supplementation are given simvastatin, a drug that decreases the activity/expression of HMG-CoA reductase, an enzyme that controls the first step of the cholesterol synthesis pathway, reduces the accumulation of toxic 7-dehydrocholesterol (immediate metabolic precursor of cholesterol) and improve neurocognitive and behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 1 years old
* Subject has confirmed diagnosis of Smith-Lemli-Opitz Syndrome
* Subject is currently receiving cholesterol supplementation

Exclusion Criteria:

* Subjects too ill to travel to the study site
* Subjects who are unable to safely undergo study procedures
* Pregnant women

Ages: 1 Year to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Roullet, PhD, Principal Investigator — Washington State University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one participant enrolled
Groups:
- Placebo - Lactose: Placebo-Lactose
  Lactose: Lactose will be administered in a capsule formula.
Period: Overall Study
Arm/Group | Placebo - Lactose | Simvastatin
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analyses were not completed and will never be completed due to insufficient funding
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Lactose | Simvastatin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Development Quotient (DQ)
Description: neurocognitive assessment measured with Mullen Scales of Learning
Time Frame: through study completion, an average of 2 per year
Population: No funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Whole Body Cholesterol Pool Size, Synthesis & Absorption Using Stable Isotope Testing
Description: administration of cholesterol and water labeled with stable isotope followed by measurement overtime in blood concentrations
Time Frame: end of treatment, an average of 1 per year
Population: Analyses were not completed and will never be completed due to insufficient funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Plasma Marker of Sterol Metabolism
Description: Blood cholesterol to 7-dehydrocholesterol ratio
Time Frame: through study completion, an average of 2 per year
Population: Analyses were not completed and will never be completed due to insufficient funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: ADC
Description: Apparent diffusion coefficient measured by brain diffusion tensor imaging (DTI)
Time Frame: end of treatment, an average of 1 per year
Population: Analyses were not completed and will never be completed due to insufficient funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: MVA
Description: urinary mevalonate excretion
Time Frame: through study completion, an average of 2 per year
Population: Analyses were not completed and will never be completed due to insufficient funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: MRS Lipids
Description: Brain magnetic resonance spectroscopy
Time Frame: end of treatment, an average of 1 per year
Population: Analyses were not completed and will never be completed due to insufficient funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: FA
Description: Fractional anisotropy as measured by brain diffusion tensor imaging (DTI)
Time Frame: end of treatment, an average of 1 per year
Population: Analyses were not completed and will never be completed due to insufficient funding
Arm/Group | Placebo - Lactose | Simvastatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Placebo - Lactose | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Analyses were not completed and will never be completed due to insufficient funding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No